CLINICAL TRIAL: NCT00185094
Title: The Effects of Olmesartan Medoxomil, Losartan Potassium, and Atenolol on Insulin Sensitivity in Overweight and Obese Subjects With Hypertension
Brief Title: A Comparison of the Effect of Olmesartan Medoxomil, Losartan Potassium, and Atenolol on the Ability of Overweight Patients With High Blood Pressure to Respond to Insulin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 866-440
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2005-12-23 (Estimated); Status verified 2005-09

CONDITIONS: Hypertension; Insulin Resistance; Metabolic Syndrome
MeSH Terms: conditions — Hypertension; Insulin Resistance; Metabolic Syndrome | interventions — Olmesartan Medoxomil; Losartan; Atenolol

INTERVENTIONS:
Drug: Olmesartan medoxomil
Drug: Losartan potassium
Drug: Atenolol

SUMMARY:
To examine the effect of three different blood pressure medications on the insulin sensitivity in overweight patients with high blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 75 years (inclusive)
* Willingness to undergo insulin clamp procedure twice
* Overweight or obese (BMI=25-39 kg/m2)
* Subject must meet one of the following two blood pressure criteria at week-2 and at week-1: Systolic blood pressure 140-179 mmHg and diastolic blood pressure 85-99 mmHg OR Systolic blood pressure < 140 mmHg and diastolic blood pressure 90-99 mmHg
* If female, must have negative serum pregnancy test at screening and be either post-menopausal, had a hysterectomy or tubal ligation at least 6 months before consent or if of childbearing potential, must practice approved measures of birth control throughout study

Exclusion Criteria:

* Systolic blood pressure > 179 mmHg
* Diastolic blood pressure > 99 mmHg or < 85 mmHg
* Diagnosis of diabetes mellitus
* History of myocardial infraction, percutaneous transluminal coronary revascularization, coronary artery bypass graft, unstable angina pectoris or an episode of heart failure requiring hospitalization
* Previous history of a cerebrovascular accident or a transient ischemic attack
* History of allergic response to atenolol, losartan potassium, olmesartan medoxomil or any of their components
* Any serious disorder, including pulmonary, hepatic, renal, gastrointestinal (including clinically significant malabsorption), uncontrolled endocrine/metabolic, hematologic/oncologic (within the last 5 years), neurologic, and psychiatric diseases, that would interfere with the conduct of the study or interpretation of the data
* Laboratory abnormalities that could compromise subject safety

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-02; Study Completion 2005-07

PRIMARY OUTCOMES:
To compare the treatment effect of olmesartan medoxomil versus that of atenolol on insulin sensitivity

SECONDARY OUTCOMES:
-To compare the treatment effect of losartan potassium versus atenolol on insulin sensitivity
-To compare the treatment effect of olmesartan medoxomil versus losartan potassium on insulin sensitivity

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Birmingham, Alabama
  - San Diego, California
  - Miami, Florida
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Rochester, Minnesota
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - San Antonio, Texas